CLINICAL TRIAL: NCT03174431
Title: A Comparison of Continence Pessary to a Disposable Intravaginal Device in the Management of Stress Urinary Incontinence: A Randomized Controlled Trial
Brief Title: Continence Pessary Versus Disposable Intravaginal Device Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Silpa Nekkanti, MD, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUI_Continence Pessary Trial
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Female Stress Incontinence

STUDY DESIGN:
Intervention Model Description: parallel group design with participants randomized to either DICD or CP (active treatment concurrent control) in a 1:1 allocation ratio for a 4-week treatment period followed by a six-month phone call follow-up to assess continued use and other treatment utilization after the initial study treatment phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continence Pessary (Active Comparator): Participants randomized to the continence pessary will be fitted for a pessary by a clinician at enrollment and they will be taught how to remove and reinsert the device. Per usual clinical practice they will be instructed to call with any concerns and scheduled for a return visit in 2 weeks for a follow-up to assess fit and comfort and undergo refitting if necessary.
  Interventions: Device: Continence Pessary
- Disposable Intravaginal Device (Active Comparator): Participants randomized to the intravaginal device will be given a sizing kit in the office, asked to select a size and provided with a 2-week supply of the appropriately sized devices. In accordance with manufacturer guidelines, participants will be instructed that the device is to be used for no more than 8 hours per 24-hour period and that each device is single use only. Participants will return in 2 weeks for a follow-up visit to assess fit and comfort, undergo resizing as necessary and receive an additional 2 week supply of the appropriately sized devices.
  Interventions: Device: Poise Impressa (Disposable Intravaginal Device)

INTERVENTIONS:
Device: Continence Pessary — Continence pessaries are inexpensive, reusable intravaginal devices made of flexible silicon that provide support to the urethra to prevent urinary leakage. Continence pessaries are fitted by trained clinicians in the office and managed by patients or their provider.
  Arms: Continence Pessary
Device: Poise Impressa (Disposable Intravaginal Device) — In 2014, the FDA approved an over-the-counter disposable intravaginal device as another nonsurgical treatment for SUI. This device is comprised of 4 support poles covered in a non-absorbable nylon mesh that is deployed using an intravaginal applicator.
  Other Names: Poise Impressa
  Arms: Disposable Intravaginal Device

SUMMARY:
This is a multi-centered randomized controlled trial of women with stress urinary incontinence or stress predominant mixed urinary incontinence who desire non-surgical therapy.

DETAILED DESCRIPTION:
In this randomized trial, eligible patients who provide written consent for participation will be enrolled. At enrollment we will collect baseline demographic data and ask participants to complete questionnaires and a 3-day bladder diary. Subjects will be randomized in a 1:1 ratio to continence pessary or disposable intravaginal device.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older (based on disposable intravaginal device manufacturing recommendations).
* SUI or SUI-predominant mixed incontinence
* English-speaking

Exclusion Criteria:

* Pregnancy
* Current symptomatic urinary tract infection (UTI).
* Postmenopausal bleeding of unknown etiology
* Neurogenic bladder
* Urinary retention (PVR >150mL obtained via bladder scan or catheterization)
* Pelvic organ prolapse past the hymen as assessed by POP-Q examination
* Inability to complete questionnaires in English or comply with study protocol
* Contraindication to pessary or disposable intravaginal device use or prior treatment or experience with either intervention.
* Prior surgery for stress urinary incontinence

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu JM, Vaughan CP, Goode PS, Redden DT, Burgio KL, Richter HE, Markland AD. Prevalence and trends of symptomatic pelvic floor disorders in U.S. women. Obstet Gynecol. 2014 Jan;123(1):141-148. doi: 10.1097/AOG.0000000000000057. PMID 24463674
- [Background] Wilson L, Brown JS, Shin GP, Luc KO, Subak LL. Annual direct cost of urinary incontinence. Obstet Gynecol. 2001 Sep;98(3):398-406. doi: 10.1016/s0029-7844(01)01464-8. PMID 11530119
- [Background] Richter HE, Burgio KL, Brubaker L, Nygaard IE, Ye W, Weidner A, Bradley CS, Handa VL, Borello-France D, Goode PS, Zyczynski H, Lukacz ES, Schaffer J, Barber M, Meikle S, Spino C; Pelvic Floor Disorders Network. Continence pessary compared with behavioral therapy or combined therapy for stress incontinence: a randomized controlled trial. Obstet Gynecol. 2010 Mar;115(3):609-617. doi: 10.1097/AOG.0b013e3181d055d4. PMID 20177294
- [Background] Ziv E, Stanton SL, Abarbanel J. Significant improvement in the quality of life in women treated with a novel disposable intravaginal device for stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jun;20(6):651-8. doi: 10.1007/s00192-009-0824-y. Epub 2009 Mar 11. PMID 19434384
- [Background] Ziv E, Stanton SL, Abarbanel J. Efficacy and safety of a novel disposable intravaginal device for treating stress urinary incontinence. Am J Obstet Gynecol. 2008 May;198(5):594.e1-7. doi: 10.1016/j.ajog.2008.01.061. Epub 2008 Apr 2. PMID 18377862
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Rogers RG, Coates KW, Kammerer-Doak D, Khalsa S, Qualls C. A short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Int Urogynecol J Pelvic Floor Dysfunct. 2003 Aug;14(3):164-8; discussion 168. doi: 10.1007/s00192-003-1063-2. Epub 2003 Jul 25. PMID 12955337
- [Background] Herzog AR, Diokno AC, Brown MB, Normolle DP, Brock BM. Two-year incidence, remission, and change patterns of urinary incontinence in noninstitutionalized older adults. J Gerontol. 1990 Mar;45(2):M67-74. doi: 10.1093/geronj/45.2.m67. PMID 2313045
- [Background] Barber MD, Kuchibhatla MN, Pieper CF, Bump RC. Psychometric evaluation of 2 comprehensive condition-specific quality of life instruments for women with pelvic floor disorders. Am J Obstet Gynecol. 2001 Dec;185(6):1388-95. doi: 10.1067/mob.2001.118659. PMID 11744914
- [Background] Meston CM. Validation of the Female Sexual Function Index (FSFI) in women with female orgasmic disorder and in women with hypoactive sexual desire disorder. J Sex Marital Ther. 2003 Jan-Feb;29(1):39-46. doi: 10.1080/713847100. PMID 12519665
- [Background] Burgio KL, Goode PS, Richter HE, Locher JL, Roth DL. Global ratings of patient satisfaction and perceptions of improvement with treatment for urinary incontinence: validation of three global patient ratings. Neurourol Urodyn. 2006;25(5):411-7. doi: 10.1002/nau.20243. PMID 16652380
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Exclusion criteria were pregnancy, current urinary tract infection (UTI), postmenopausal bleeding, neurogenic bladder, urinary retention, pelvic organ prolapse past the hymen, contraindication to device use, prior treatment with either device, and prior surgery for SUI. Women excluded for a current symptomatic UTI were eligible for enrollment after treatment was completed and a negative urine culture was obtained.
Period: Overall Study
Arm/Group | Continence Pessary | Disposable Intravaginal Device
Started | 25 | 25
Completed | 8 | 9
Not Completed | 17 | 16
Not completed — Withdrawal by Subject | 14 | 11
Not completed — alternative treatment | 2 | 0
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continence Pessary | Disposable Intravaginal Device | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [43 to 52] | 41 [38 to 49] | 44 [40 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success
Description: Success of stress urinary incontinence treatment is defined as a response of "very much better" or "much better" on the Patient Global Impression of Improvement (PGI-I).
Time Frame: 4 weeks
Population: Discrepancy in analyzed numbers is secondary to patients either withdrawing from study, lost to follow up, or choosing alternative treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Continence Pessary | Disposable Intravaginal Device
Number analyzed (Participants) | 10 | 12
Participants | 8 | 9

2. Secondary Outcome: Validated Questionnaires
Description: Validated questionnaire scores obtained at baseline and week 4 with all questionnaires having higher scores indicating higher level of bother:
  1. Urinary Distress Inventory (UDI-6): 6 questions measuring urinary incontinence symptom bother. Scale: 0-600.
  2. Incontinence Impact Questionnaire (IIQ-7): 7 questions measuring functional impact of urinary incontinence. Scale: 0-100.
  3. Female Sexual Function Index (FSFI) : 19 items use a 5-point Likert scale (1-5) to assess sexual functioning in women in 6 domains (Desire, arousal, lubrication, orgasm, satisfaction, pain). Sum of each domain is multiplied by a factor ratio (0.6: desire; 0.3: arousal and lubrication; 0.4: orgasm, satisfaction, and pain) to have all domain totals on a comparable scale.
  Score ranges for each domain:
  1. Desire: 1.2- 6
  2. Arousal, lubrication, orgasm, and pain: 0- 6
  3. Satisfaction: 0.8- 6 They are then summed to derive a total FSFI score of 2- 36.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continence Pessary | Disposable Intravaginal Device
Number analyzed (Participants) | 10 | 12
score on a scale
  UDI-6 | 110 (135) | 71 (105)
  IIQ-7 | 10 (30) | 7 (12)
  FSFI | -1 (0) | 1 (2)

3. Secondary Outcome: Satisfaction With Device
Description: Satisfaction with device will be assessed using likert scale questionnaires assessing device satisfaction, ease of use, comfort, and likelihood of continued use at 4 weeks.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Continence Pessary | Disposable Intravaginal Device
Number analyzed (Participants) | 10 | 12
participants
  Satisfied with device | 5 | 4
  Device is comfortable | 7 | 10
  Device is easy to use | 8 | 12
  High likely to continue using | 8 | 7

4. Secondary Outcome: Adverse Events
Description: Potential adverse events of interest include vaginal discomfort, vaginal bleeding, vaginal infection, vaginal abrasion/laceration, and urinary tract infection (UTI)
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Continence Pessary | Disposable Intravaginal Device
Number analyzed (Participants) | 10 | 12
Participants | 1 | 0

5. Secondary Outcome: 6 Month Follow up
Description: 6 month intervention use and satisfaction with following questions as yes or no:
  1. Still using device
  2. Using other SUI treatment ( pessary, physical therapy)
  3. Satisfied with treatment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Continence Pessary | Disposable Intravaginal Device
Number analyzed (Participants) | 8 | 9
Participants
  Still using device | 5 | 4
  Using Pessary | 0 | 2
  Physical therapy | 0 | 1
  Satisfied with treatment | 4 | 5

ADVERSE EVENTS:
Time Frame: 6 months from completion of study.
Description: There were no serious adverse events in the study. Only one adverse event occurred, a patient randomized to continence pessary removed the device after the fitting visit because of discomfort. She was treated with vaginal estrogen and was refit.
Arm/Group | Continence Pessary | Disposable Intravaginal Device
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 0/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continence Pessary (N=25) | Disposable Intravaginal Device (N=25)
Vaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT03174431/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT03174431/ICF_001.pdf